CLINICAL TRIAL: NCT06035341
Title: Is There a Association Between Temporomandibular Disorders and Sacroiliac Joint Dysfunction?
Brief Title: The Association Between Temporomandibular Disorders and Sacroiliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2023.675
Record Dates: First submitted 2023-08-25; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Disorder
Keywords: Temporomandibular Joint Disorders; Temporomandibular Joint; Sacroiliac Joint; Orofacial Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Intervention Model Description: There are one study group. A single session of orofacial manual therapy will be applied to all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Participants in this group will be received orofacial manual therapy as treatment. The number of participants is planned to be 23.
  Interventions: Other: Orofacial Manual Therapy

INTERVENTIONS:
Other: Orofacial Manual Therapy — As orofacial manual therapy, soft tissue (intraoral and extraoral trigger point therapy and myofascial release of painful muscles) and joint mobilization (caudal and ventro-caudal traction, ventral and mediolateral translation), muscle energy technique, fascia mandibularis release, occipital release and ligamentous treatment was planned.

SUMMARY:
The aim of this study is to evaluate the relationship between Temporomandibular Disorders (TMD) and Sacroiliac Joint Disfunction (SIJD) and to determine the immediate effect of single-session orofacial manual therapy on SIJD. Patients will be treated for 1 session. The evaluation was planned to be done twice, at the beginning and end of the session.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the relationship between TMD and SIJD and to determine the immediate effect of single-session orofacial manual therapy on SIJD. Patients diagnosed with both TMD and SIJD will be participants of the study. Patients will be treated for 1 session. Immediately after the treatment, participants will be asked to walk for 5 minutes, after which a second assessment will be done. The evaluation was planned to be done twice, at the beginning and end of the session. Pressure pain threshold, joint range of motion, functionality, and sacroiliac joint disfunction will be evaluated by using digital algometer, ruler, "Oswestry Disability Index (ODI)" and specific tests respectively.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate,
* Aged between 18-60 years old,
* Having the diagnosis of Temporomandibular Disorders (TMB) and sacroiliac joint disfunction (SIJD),

Exclusion Criteria:

* Having a malignant condition, trauma and surgery of the cranial and cervical region,
* Not being cooperative,
* Regular use of analgesic and anti-inflammatory drugs,
* Having dentofacial anomalies,
* Having active inflammatory arthritis,
* Having metabolic diseases (Gout, osteoporosis, Cushing's disease and hyper/hypo-parathyroidism),
* Having connective tissue, rheumatological (Systemic lupus erythematosus and scleroderma) and hematological disorders (Anemia and leukemia),
* Having a diagnosed psychiatric illness,
* Receiving TMD-related physical therapy less than 6 months ago

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Pain Threshold: Digital algometer | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  The algometer is a reliable instrument for measuring the sensitivity of the masticatory muscles and 1 cm below the Posterior Superior Iliac Spine (PSIS). The measurement will be made at 10 points. A force (Newton in force) of 1 kg (weight in kilogram) per square centimeter (surface area in centimeter square) is applied to the patient for 3 seconds, and this is continued until the patient feels pain (weight and surface area will be combined to report Newton in kg/ cm2). This process will be repeated three times and the average value will be calculated.
Range of Motion | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  Mouth opening, protrusion and right and left lateral deviation will be measured starting from 0 using a 15 cm ruler. Repeated measuring reduces the standard error of measurement, hence repeated measurements will be also included in our study (three times) with the largest recorded range taken.
First Test for Sacroiliac Joint Disfunction: Distraction Test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  The patient lies in a supine position. Direct posterolateral pressure is applied to the bilateral anterior superior iliac spines, thus stressing the anterior sacroiliac ligament. Pathology in the Sacroiliac (SI) joint is considered if pain occurs in the hip.
Second Test for Sacroiliac Joint Disfunction: Compression Test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  The patient lies on his side with the affected side on top, with the hip at 45° flexion and the knees at 90° flexion. The physician stands behind the patient and applies pressure to the pelvis over the iliac crest directly toward the contralateral iliac crest. This test can be applied in a supine or prone position. Pathology in the SI joint is considered if pain occurs in the hip.
Third Test for Sacroiliac Joint Disfunction: Thigh Thrust Test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  The patient lies in a supine position. The hip is brought to 90º flexion. Pressure is applied directly toward the examination table. Pathology in the SI joint is considered if pain occurs in the hip. Pain provocation is established with hip flexion and adduction.
Fourth Test for Sacroiliac Joint Disfunction: Gaenslen Test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  The patient lies in a supine position close to the edge of the bed. The patient draws his leg toward the abdomen so as to place the knee and hip in flexion. The outside leg (closest to the practitioner) is allowed to hang down from the examination table, while the SI joint is contracted by placing pressure on the inside (furthest from the practitioner) iliac crest and outside leg. Pain indicates pathology of the SI joint on the tested side.
Fifth Test for Sacroiliac Joint Disfunction: Sacral Thrust Test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  The patient lies in a prone position. The practitioner places one hand on the apex of the sacrum while applying direct pressure with the other hand. Pathology in the SI joint is considered if pain occurs in the hip.
Sixth Test for Sacroiliac Joint Disfunction: Faber (Patrick) Test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). The intervention is one hour.
  The patient lies in a supine position, while the practitioner stands beside the patient and bends the patient's knee, bringing the heel to the opposite knee. With the other hand, the practitioner ensures that the contralateral anterior superior iliac spine remains in a neutral position. The physician applies mild pressure to the bent knee. Pressure is assumed to be applied to the bilateral SI ligaments and hip joints. Pathology in the SI joint is considered if pain occurs in the hip. Pain provocation occurs with flexion, adduction and external rotation of the hip.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) for Functional Low Back Pain | Change between baseline (immediately before intervention) and 1 week post intervention. The intervention is one hour.
  Oswestry Disability Index (ODI) will be used to evaluate low back pain. ODI consists of 10 items on the degree of severity to which low back trouble has affected the ability to manage in everyday life. The 10 sections cover the pain and the daily function (including pain intensity, personal hygiene, lifting, walking, sitting, standing, sleeping, sexual activity, social activity, and traveling). Each item is rated on a 6-point scale (0-5); the higher score means the higher level of disability related to low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Kuru Colak, Asst. Prof, Study Director — Marmara University Institute of Health Sciences
Locations (1):
- Sultan İğrek, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) might be considered to be shared with clinicians studying in the same field one year after the publication of the study.

REFERENCES:
- [Background] Anastassaki Kohler A, Hugoson A, Magnusson T. Prevalence of symptoms indicative of temporomandibular disorders in adults: cross-sectional epidemiological investigations covering two decades. Acta Odontol Scand. 2012 May;70(3):213-23. doi: 10.3109/00016357.2011.634832. Epub 2011 Nov 30. PMID 22126531
- [Background] Kiapour A, Joukar A, Elgafy H, Erbulut DU, Agarwal AK, Goel VK. Biomechanics of the Sacroiliac Joint: Anatomy, Function, Biomechanics, Sexual Dimorphism, and Causes of Pain. Int J Spine Surg. 2020 Feb 10;14(Suppl 1):3-13. doi: 10.14444/6077. eCollection 2020 Feb. PMID 32123652
- [Background] Gregory TM. Temporomandibular disorder associated with sacroiliac sprain. J Manipulative Physiol Ther. 1993 May;16(4):256-65. PMID 8340721
- [Background] Chinappi AS Jr, Getzoff H. Chiropractic/dental cotreatment of lumbosacral pain with temporomandibular joint involvement. J Manipulative Physiol Ther. 1996 Nov-Dec;19(9):607-12. PMID 8976480
- [Background] Fink M, Wahling K, Stiesch-Scholz M, Tschernitschek H. The functional relationship between the craniomandibular system, cervical spine, and the sacroiliac joint: a preliminary investigation. Cranio. 2003 Jul;21(3):202-8. doi: 10.1080/08869634.2003.11746252. PMID 12889677
- [Background] Tuncer AB, Ergun N, Tuncer AH, Karahan S. Effectiveness of manual therapy and home physical therapy in patients with temporomandibular disorders: A randomized controlled trial. J Bodyw Mov Ther. 2013 Jul;17(3):302-8. doi: 10.1016/j.jbmt.2012.10.006. Epub 2012 Nov 16. PMID 23768273
- [Background] Kalamir A, Pollard H, Vitiello A, Bonello R. Intra-oral myofascial therapy for chronic myogenous temporomandibular disorders: a randomized, controlled pilot study. J Man Manip Ther. 2010 Sep;18(3):139-46. doi: 10.1179/106698110X12640740712374. PMID 21886424
- [Background] von Piekartz H, Ludtke K. Effect of treatment of temporomandibular disorders (TMD) in patients with cervicogenic headache: a single-blind, randomized controlled study. Cranio. 2011 Jan;29(1):43-56. doi: 10.1179/crn.2011.008. PMID 21370769
- [Background] Walker N, Bohannon RW, Cameron D. Discriminant validity of temporomandibular joint range of motion measurements obtained with a ruler. J Orthop Sports Phys Ther. 2000 Aug;30(8):484-92. doi: 10.2519/jospt.2000.30.8.484. PMID 10949505
- [Background] Telli H, Telli S, Topal M. The Validity and Reliability of Provocation Tests in the Diagnosis of Sacroiliac Joint Dysfunction. Pain Physician. 2018 Jul;21(4):E367-E376. PMID 30045603
- [Background] Robinson HS, Brox JI, Robinson R, Bjelland E, Solem S, Telje T. The reliability of selected motion- and pain provocation tests for the sacroiliac joint. Man Ther. 2007 Feb;12(1):72-9. doi: 10.1016/j.math.2005.09.004. Epub 2006 Jul 12. PMID 16843031
- [Background] Laslett M, Young SB, Aprill CN, McDonald B. Diagnosing painful sacroiliac joints: A validity study of a McKenzie evaluation and sacroiliac provocation tests. Aust J Physiother. 2003;49(2):89-97. doi: 10.1016/s0004-9514(14)60125-2. PMID 12775204
- [Background] Martin RL, Sekiya JK. The interrater reliability of 4 clinical tests used to assess individuals with musculoskeletal hip pain. J Orthop Sports Phys Ther. 2008 Feb;38(2):71-7. doi: 10.2519/jospt.2008.2677. Epub 2007 Sep 21. PMID 18560194
- [Background] Cattley P, Winyard J, Trevaskis J, Eaton S. Validity and reliability of clinical tests for the sacroiliac joint. A review of literature. Australas Chiropr Osteopathy. 2002 Nov;10(2):73-80. PMID 17987177
- [Background] Laslett M, Aprill CN, McDonald B, Young SB. Diagnosis of sacroiliac joint pain: validity of individual provocation tests and composites of tests. Man Ther. 2005 Aug;10(3):207-18. doi: 10.1016/j.math.2005.01.003. PMID 16038856
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- See also: Investigation of the Relationship Between Temporomandibular Disorder and Postural Analysis — https://jag.journalagent.com/kocaelitip/pdfs/KTD_10_2_27_32.pdf
- See also: Manual Therapy for Temporomandibular Disorders: A Review of the Literature. — https://www.semanticscholar.org/paper/Manual-therapy-for-temporomandibular-disorders%3A-A-Kalamir-Pollard/eff17b74aec032c4f05e66879a61cd158ddda70d
- See also: Pressure Pain Threshold and Pain Perception in Temporomandibular Disorder Patients: Is There Any Correlation? — https://www.scielo.br/j/rdor/a/dV5P7vngMkggzjZqKrCvHsR/?lang=en